CLINICAL TRIAL: NCT06624163
Title: Evaluation of Patient Coach Support for Older Adults With Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shenbagam Dewar, Clinical Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00210504; P30AG024824 (NIH)
Record Dates: First submitted 2024-09-26; First posted 2024-10-02 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Health Coach; Aging
MeSH Terms: conditions — Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental)
  Interventions: Behavioral: OHWL Clinic Activities (Standard of Care); Behavioral: Coach Activities

INTERVENTIONS:
Behavioral: OHWL Clinic Activities (Standard of Care) — Following a directed history and physical at the initial visit, the OHWL Care provider (OCP) develops a medical and weight management plan, which includes laboratory testing (such as for Hemoglobin A1C (HbA1c), consultant referrals (e.g. sleep, heart failure clinics) and referral to nutritionists and physical therapy (PT). The OCP begins the process of establishing patient goals, which will be followed up by the coach. The OCP reviews patient progress with the goals during face-to-face visits (some by telehealth) at two, four and six months. As part of the standard initial clinic evaluation, a medical assistant evaluates grip strength (using a hand dynamometer) the timed up and go mobility test; these are repeated at the 6-month visit.
Behavioral: Coach Activities — A patient coach follows patients outside of clinic to ensure adherence with referral appointments and use of recommended community services. The coach assesses the participant at baseline, 3 months, and 6 months using the Patient-Specific Functional Scale and follows up with patients via phone over 6 months. The coach utilizes S.M.A.R.T. (Specific, Measurable, Achievable, Relevant, Time-bound) goals to facilitate, for example, transportation, barriers to scheduling, etc. The coach follows up on specialist referral recommendations, physical therapy, and nutrition program, as well as social work recommendations. Barriers and facilitators to program adherence are identified and addressed.

SUMMARY:
The purpose of the present pilot is to evaluate the outcomes of adding a patient coach to support the Optimal Health Weight and Lifestyle (OHWL) Clinic plan developed by PI Dewar, specifically to address barriers and facilitators of adherence to the plan. This will be accomplished via a coach who is not embedded in clinic care and is supported by pilot research funds. Evaluation of the coach activities, conducted by research personnel, will include compiling data from the electronic health record, a short set of patient report and performance measures, and qualitative interviews.

DETAILED DESCRIPTION:
A patient coach added to the OHWL Clinic plan as part of the pilot will help patients who are being treated for weight loss to achieve their goals, help address barriers and facilitators of adherence to referred services such physical therapy and nutritionist appointments and various specialists and links to community services as needed. Evaluation of the coach activities will be conducted by research personnel, which will also include data compilation from the electronic health record, a short set of patient report and performance measures, and qualitative interviews. This project will provide pilot data for future funding proposals.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) equal to or greater than 35
* Ability to walk across a room with or without an assistive device
* Willingness and ability to follow instructions
* Interest in weight management
* At least two of the following conditions: hypertension, cardiovascular conditions including heart failure, diabetes mellitus, hyperlipidemia, non-alcoholic steatohepatitis, obstructive sleep apnea, osteoarthritis

Exclusion Criteria:

* Active mental health disorder, such as major depression
* Moderate to severe cognitive impairment
* Mobility limited to bed-bound status

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who attend physical therapy appointments | 6 months
  Patients who reported attending at least one physical therapy appointment during the course of the study, if referred.
Percentage of participants who achieve treatment goals | 6 months
  Percentage of participants whose coaches reported successful achievement of established goals for diet and physical therapy based on end of study interview.
Percentage of participants who attend nutritional consultation appointments | 6 months
  Patients who reported attending at least one nutritional consultation appointment during the course of the study.
Percentage of participants who access community resources | 6 months
  Patients who reported using a community resource (such as a gym, community park, or other similar resource) at least once during the course of the study.

SECONDARY OUTCOMES:
Change in PROMIS-29 Score (Patient-Reported Outcomes Measurement Information System) | 6 months
  PROMIS 29 questionnaire gauges health-related quality of life across seven key domains: physical function, pain interference, fatigue, sleep disturbance, physical and mental health, and social health. Each item is auto-scored and T-score is obtained for each domain and will be tracked during the study time frame
  Scores range from 0 to 100, where a score of 0 indicates lowest quality of life and 100 indicates highest quality of life.
Change in reported participant pain levels | 6 months
  This is assessed by PROMIS-Global Pain instrument which is a survey administered to patient by Computer adaptive testing, Scale 0-10 (where 0 is no pain and 10 is worst pain imaginable) and will track change during study period
Change in NHATS (National health and aging trends study) Score | 6 months
  NHATS instrument scores individual's self-report of difficulty or dependency with performing activities of daily living such as self-care and mobility and restrictions in instrumental activities of daily living domains. Each domain has multiple questions with responses such as (Yes/No) for most; (None, little, some, Lot); (Always did it by self, together with someone else, someone always did it, it varied, not done in the last month); (everyday, most days, some days, rarely, never); (every time, most times, sometimes, rarely).
Change in patient mobility | 6 months, 12 months
  Mobility and balance is measured during clinic visits using TUG (Timed up and go). The patient is asked to rise from a seated position, walk 3 m, turn around, and return and sit in the starting point chair while timed. Patients who fail to complete the test in fewer than 12 s are considered to have elevated fall risk Measurements will be taken every six months.
Change in Life Space Assessment Score | 6 months
  Life-space mobility is a measure of resilience to physical decline and social isolation in older adults. They are nine 'yes/no' questions regarding a person's movements across nine life-space zones in the preceding 3 days. The total score ranges from 0 to 9, where 0 means most restricted life-space and 9 is least restricted life-space.

OTHER OUTCOMES:
NUTRITION assessment by ASA24 food recall - fat | 6 months
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls. Participants are asked to report everything they ate or drank over the last 24-hours by using an online tool. Data collected on enrollment and 3 months and at 6 months. Intake of grams fat will be tracked to see changes over the study period.
NUTRITION assessment by ASA24 food recall - kilocalories | 6 months
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls. Participants are asked to report everything they ate or drank over the last 24-hours by using an online tool. Data collected on enrollment and 3 months and at 6 months. Intake of total kilocalories will be tracked to see changes over the study period.
NUTRITION assessment by ASA24 food recall - saturated fat | 6 months
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls. Participants are asked to report everything they ate or drank over the last 24-hours by using an online tool. Data collected on enrollment and 3 months and at 6 months. Intake of grams saturated fat will be tracked to see changes over the study period.
NUTRITION assessment by ASA24 food recall - sodium | 6 months
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls. Participants are asked to report everything they ate or drank over the last 24-hours by using an online tool. Data collected on enrollment and 3 months and at 6 months. Intake of milligrams sodium will be tracked to see changes over the study period.
NUTRITION assessment by ASA24 food recall - added sugar | 6 months
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls. Participants are asked to report everything they ate or drank over the last 24-hours by using an online tool. Data collected on enrollment and 3 months and at 6 months. Intake of grams of added sugar will be tracked to see changes over the study period.
NUTRITION assessment by ASA24 food recall - alcohol | 6 months
  The Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool is a web-based tool that enables multiple, automatically coded self-administered 24-hour recalls. Participants are asked to report everything they ate or drank over the last 24-hours by using an online tool. Data collected on enrollment and 3 months and at 6 months. Intake of grams of alcohol will be tracked to see changes over the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan - East Ann Arbor Geriatrics Center, Ann Arbor, Michigan, United States